CLINICAL TRIAL: NCT02446457
Title: Phase II Study of Rituximab Plus Pembrolizumab (MK-3475) in Subjects With Relapsed Follicular Lymphoma
Brief Title: Rituximab and Pembrolizumab With or Without Lenalidomide in Treating Patients With Relapsed Follicular Lymphoma and Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0539; NCI-2015-01307 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0539 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Lenalidomide; pembrolizumab; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (rituximab, pembrolizumab) (Experimental): Patients receive rituximab IV over 4-8 hours on days 1, 8, 15, and 22. Patients also receive pembrolizumab IV over 1 hour on day 2 every 3 weeks for up to 16 cycles (1 year) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Biological: Rituximab
- Cohort II (rituximab, pembrolizumab, lenalidomide) (Experimental): Patients receive rituximab IV over 4-8 hours on days 1, 8 and 15 of cycle 1, and day 1 of cycle 2. Patients also receive pembrolizumab IV over 1 hour on day 2 every 3 weeks for up to 2 years, and lenalidomide PO on days 1-14 every 3 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Pembrolizumab; Biological: Rituximab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
  Arms: Cohort II (rituximab, pembrolizumab, lenalidomide)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies how well rituximab and pembrolizumab with or without lenalidomide works in treating patients with follicular lymphoma and diffuse large B-cell lymphoma that has returned after a period of improvement. Immunotherapy with monoclonal antibodies, such as rituximab and pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving rutuximab with pembrolizumab and lenalidomide may work better at treating follicular lymphoma and diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) in subjects with relapsed follicular lymphoma (FL) treated with rituximab plus pembrolizumab.

II. To determine the ORR in subjects with relapsed/refractory FL and relapsed/refractory diffuse large B-cell lymphoma (DLBCL) who have failed chimeric antigen receptor (CAR) T cell therapy and are treated with rituximab in combination with pembrolizumab and lenalidomide. (Cohort 2)

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity. II. To determine the complete response rate (CRR). III. To determine the overall progression-free survival (PFS). IV. To compare PFS between patients relapsing =< one year vs > one year after last prior therapy.

V. To determine the overall survival (OS). VI. To determine the safety and toxicity. (Cohort 2) VII. To determine the CRR. (Cohort 2) VIII. To determine the overall PFS. (Cohort 2) IX. To compare PFS between patients relapsing =< one year vs > one year after last prior therapy. (Cohort 2) X. To determine the OS. (Cohort 2)

EXPLORATORY OBJECTIVES:

I. To determine effects of rituximab plus pembrolizumab therapy on peripheral blood T cells.

II. To correlate features of peripheral blood T cells with toxicities after rituximab plus pembrolizumab therapy.

III. To correlate features of peripheral blood T cells with response and PFS after rituximab plus pembrolizumab therapy.

IV. To correlate baseline tumor characteristics with response and PFS after rituximab plus pembrolizumab therapy.

V. To determine effects of rituximab, pembrolizumab, and lenalidomide therapy on peripheral blood T cells. (Cohort 2) VI. To correlate features of peripheral blood T cells with toxicities after rituximab, pembrolizumab, and lenalidomide therapy. (Cohort 2) VII. To correlate features of peripheral blood T cells with response and PFS after rituximab, pembrolizumab, and lenalidomide therapy. (Cohort 2) VIII. To correlate baseline tumor characteristics with response and PFS after rituximab, pembrolizumab, and lenalidomide therapy. (Cohort 2)

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive rituximab intravenously (IV) over 4-8 hours on days 1, 8, 15, and 22. Patients also receive pembrolizumab IV over 1 hour on day 2 every 3 weeks for up to 16 cycles (1 year) in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive rituximab IV over 4-8 hours on days 1, 8 and 15 of cycle 1, and day 1 of cycle 2. Patients also receive pembrolizumab IV over 1 hour on day 2 every 3 weeks for up to 2 years, and lenalidomide orally (PO) on days 1-14 every 3 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* For cohort 1: Male or female subjects with histologic proof of follicular lymphoma grade 1, 2, or 3a relapsing after at least one prior systemic therapy that included rituximab (or other monoclonal CD20 antibody); patients should have documented rituximab-sensitive disease defined as a documented complete or partial response lasting at least 6 months after the last rituximab-containing therapy
* For cohort 2: Male or female subjects with histologic proof of follicular lymphoma grade 1, 2, or 3a relapsing after at least two prior systemic therapies, which must include CAR T cell therapy or histologic proof of DLBCL relapsing after at least two prior systemic therapies, which must include CAR T cell therapy
* Either the subject or his/her legally authorized representative be willing and able to provide written informed consent for the trial
* Have measurable disease (>= 1.5 cm in the longest diameter for nodal or extranodal disease)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L, performed within 28 days of treatment initiation
* Platelets >= 50 x 10^9/L, performed within 28 days of treatment initiation
* Hemoglobin >= 8.0 g/dL, performed within 28 days of treatment initiation
* Serum creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min GFR or CrCl for subjects with creatinine levels > 1.5 x institutional ULN, performed within 28 days of treatment initiation

  * Creatinine clearance will be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN, performed within 28 days of treatment initiation
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) =< 2.5 x ULN OR =< 5 x ULN for subjects with lymphoma in the liver, performed within 28 days of treatment initiation
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants performed within 28 days of treatment initiation
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants, performed within 28 days of treatment initiation
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; female subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

  * Females of reproductive potential enrolled in the lenalidomide cohort must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Male subjects should agree to use two methods of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* All study participants enrolled in the lenalidomide containing cohort (cohort 2) must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study drug or using an investigation device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from AEs due to a previously administered agent; * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing and requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) lymphoma and/or lymphomatous meningitis; subjects with previously treated CNS lymphoma and/or lymphomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* No active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators, local steroid injections or inhaled or topical steroids would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), anti-programmed cell death ligand 2 (PD-L2), anti- cluster of differentiation (CD)137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)

  * Note: Subjects that received prior therapy with pidilizumab are an exception to this criterion and may qualify for the study
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] qualitative is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (complete + partial responses) | Up to 2 years after completion of study treatment
  Overall response will be monitored simultaneously using the Bayesian stopping boundaries calculated based on beta-binomial distributions. Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate.

SECONDARY OUTCOMES:
Incidence of toxicity | Up to 30 days after the completion of study treatment
  Will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Toxicity will be monitored simultaneously using the Bayesian stopping boundaries calculated based on beta-binomial distributions. Toxicity defined as any grade 3 or 4 non-hematologic toxicity that in the opinion of the principal investigator is at least possibly related to study treatment. Toxicity evaluation will be based on the incidence of severity and type of adverse events (including physical and laboratory). Frequency tables will be used to summarize categorical variables. Logistic regression will be utilized to assess the effect of patient prognostic factors on the toxicity rate.
Complete response rate | Up to 2 years after completion of study treatment
  Logistic regression will be utilized to assess the effect of patient prognostic factors on the response rate.
Progression-free survival (PFS) | Up to 2 years after completion of study treatment
  The PFS will be compared between patients relapsing =< 1 year vs > 1 year after last prior therapy. The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.
Overall survival | Up to 2 years after completion of study treatment
  The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test. Cox proportional hazard regression will be employed for multivariate analysis on time-to-event outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Nair, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Nastoupil LJ, Chin CK, Westin JR, Fowler NH, Samaniego F, Cheng X, Ma MCJ, Wang Z, Chu F, Dsouza L, Obi C, Mims J, Feng L, Zhou S, Green M, Davis RE, Neelapu SS. Safety and activity of pembrolizumab in combination with rituximab in relapsed or refractory follicular lymphoma. Blood Adv. 2022 Feb 22;6(4):1143-1151. doi: 10.1182/bloodadvances.2021006240. PMID 35015819
- See also: M D Anderson Cancer Center — http://www.mdanderson.org